CLINICAL TRIAL: NCT01077284
Title: A Multicenter, Randomized, Double-Blind, Placebo and Allopurinol Controlled, Phase 2 Study to Evaluate Febuxostat in the Medical Management of Subjects With Hyperuricosuria and Calcium Oxalate Stones
Brief Title: Febuxostat Versus Allopurinol or Placebo in Patients With Hyperuricosuria and Calcium Oxalate Stones
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMX-67_201; U1111-1113-6322 (Registry Identifier: WHO)
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-01

CONDITIONS: Hyperuricosuria; Kidney Stones
Keywords: Kidney Calculi; Kidney Stones; Nephrolithiasis; Drug Therapy; Uric Acid
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis | interventions — Febuxostat; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Febuxostat (Experimental): Febuxostat 80 mg, capsules, orally, once daily for up to 6 months.
  Interventions: Drug: Febuxostat
- Allopurinol (Active Comparator): Allopurinol 200mg or 300mg (determined by kidney function), capsules, orally, once daily for up to 6 months.
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): Placebo-matching capsules, orally, once daily for up to 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Febuxostat — Febuxostat capsules
  Other Names: Uloric; TMX-67
  Arms: Febuxostat
Drug: Allopurinol — Allopurinol capsules
  Other Names: Zyloprim
  Arms: Allopurinol
Drug: Placebo — Placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of febuxostat, once daily (QD), compared to allopurinol or placebo in patients with excessive amounts of uric acid in their urine and who have recently had kidney stones.

DETAILED DESCRIPTION:
Nephrolithiasis, also called kidney stone disease, occurs in patients with genetic susceptibility and who may have a broad spectrum of metabolic disorders and other comorbid conditions (for example obesity or diabetes). These renal stones develop as a result of supersaturation. Calcium oxalate (CaOx) is the most common type of stone. Reducing the urinary excretion of uric acid is an established approach for the treatment of CaOx kidney stones.

The objective of this study is to evaluate treatment with febuxostat compared to allopurinol or placebo in the reduction of 24-hour urine uric acid (uUA) excretion levels in hyperuricosuric patients with a recent history of renal stones and the presence of at least one CaOx stone larger than or equal to 3 mm as seen on Multidetector Computed Tomographic Angiography (MDCT).

Participants in this study will be required to make 4 office visits provide 3 urine samples and undergo 2 MDCT scans (a type of x-ray) of their kidneys.

ELIGIBILITY:
Inclusion Criteria:

* Has hyperuricosuria, defined as a daily urine uric acid excretion greater than 700 mg as measured by 24-hour urine collection prior to randomization.
* Has at least one calcium oxalate stone greater than or equal to 3 mm in its longest in-plane diameter, identified by Multiple Detector Computated Tomography prior to randomization.
* Has a recent (within the previous 5 years) history of renal stones prior to screening.

Exclusion Criteria:

* Has gout, secondary hyperuricemia or has experienced a gout flare.
* Has a history of xanthinuria.
* Has received allopurinol or probenecid within 2 years prior to randomization.
* Has received febuxostat.
* Has alanine aminotransferase and/or aspartate aminotransferase values greater than 2.0 times the upper limit of normal at the Screening Visit.
* Has an abnormal serum calcium level at the Screening Visit.
* Has a significant medical condition and/or conditions that would interfere with the treatment, safety or compliance with the protocol according to the judgment of the Investigator.
* Has a history of drug abuse or a history of alcohol abuse within 5 years prior to the Screening Visit.
* Participant's measured creatinine clearance is less than 30 mL/min at the Screening Visit.
* Has hypercalciuria at Screening, while on a regular unrestricted diet, defined as urinary excretion of:

  * greater than 250 mg of calcium/24-hour for females of body weight less than 62.5 kg; OR
  * greater than 300 mg calcium/24-hour for males of body weight less than 75 kg; OR
  * greater than 4 mg calcium/kg/24-hour for males of body weight greater than or equal 75 kg and females of body weight greater than or equal 62.5 kg.

EXCLUDED MEDICATIONS:

* Febuxostat, allopurinol, probenecid.
* Salicylates (chronic use of aspirin ≤325 mg/day is allowed).
* Azathioprine.
* Mercaptopurine.
* Theophylline.
* Colchicine.
* Pyrazinamide.
* Sulfamethoxazole/trimethoprim.
* Losartan.

The following restrictions also apply during the study:

* Long-term use (more than 4 continuous weeks) of prescription or over-the-counter nonsterioidal anti-inflammatory drugs or cyclooxygenase-2 inhibitors.
* If receiving diuretics, participant must have been on a stable dose for at least 30 days prior to screening. No changes in dosage are allowed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director Clinical Science, Study Director — Takeda
Locations (28):
- United States (28):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Tucson, Arizona
  - Costa Mesa, California
  - Orange, California
  - Palmdale, California
  - Poway, California
  - Rancho Cucamonga, California
  - San Diego, California
  - Santa Ana, California
  - Denver, Colorado
  - New Britain, Connecticut
  - Miami, Florida
  - Augusta, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Meridian, Idaho
  - Lexington, Kentucky
  - Kalamazoo, Michigan
  - Jackson, Mississippi
  - Albuquerque, New Mexico
  - New Windsor, New York
  - Shelby, North Carolina
  - Wilmington, North Carolina
  - East Providence, Rhode Island
  - Dallas, Texas
  - Houston, Texas
  - Sugar Land, Texas

REFERENCES:
- [Derived] Goldfarb DS, MacDonald PA, Gunawardhana L, Chefo S, McLean L. Randomized controlled trial of febuxostat versus allopurinol or placebo in individuals with higher urinary uric acid excretion and calcium stones. Clin J Am Soc Nephrol. 2013 Nov;8(11):1960-7. doi: 10.2215/CJN.01760213. Epub 2013 Aug 8. PMID 23929928
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 24 investigative sites in the United States from 12 February 2010 to 21 November 2011.
Pre-assignment Details: Participants with hyperuricosuria and calcium oxalate stones were randomized to 1 of 3 treatment groups in a 1:1:1 ratio to receive placebo, allopurinol or febuxostat.
Period: Overall Study
Arm/Group | Febuxostat | Allopurinol | Placebo
Started | 33 | 33 | 33
Completed | 28 | 28 | 30
Not Completed | 5 | 5 | 3
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 1
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat | Allopurinol | Placebo | Total
Number analyzed (Participants) | 33 | 33 | 33 | 99
Age Continuous [Mean (Standard Deviation); unit: years] | 49.1 (9.69) | 46.5 (9.95) | 46.5 (11.54) | 47.4 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 6 | 14
  Male | 27 | 31 | 27 | 85
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 8 | 8 | 3 | 19
  Non-Hispanic and Latino | 25 | 25 | 30 | 80
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 0 | 2 | 4
  Black or African American | 3 | 1 | 1 | 5
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1 | 2
  White | 26 | 31 | 29 | 86
  Other | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 33 | 99
Height [Mean (Standard Deviation); unit: cm] | 172.6 (12.67) | 176.5 (7.71) | 174.3 (9.31) | 174.5 (10.14)
Weight [Mean (Standard Deviation); unit: kg] | 98.0 (18.17) | 100.9 (20.13) | 100.8 (20.23) | 99.9 (19.38)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.9 (5.71) | 32.3 (5.82) | 33.1 (6.29) | 32.8 (5.89)
Body mass index categories [Number; unit: participants]
  18.5 to <25 kg/m^2 | 2 | 1 | 2 | 5
  25 to <30 kg/m^2 | 8 | 14 | 7 | 29
  ≥30 kg/m^2 | 23 | 18 | 24 | 65
Baseline Serum Urate [Mean (Standard Deviation); unit: mg/dL] | 6.2 (1.63) | 6.3 (1.49) | 6.3 (1.24) | 6.3 (1.45)
Baseline Serum Urate categories [Number; unit: participants]
  <9.0 mg/dL | 31 | 31 | 32 | 94
  9.0 to <10 mg/dL | 2 | 0 | 1 | 3
  ≥10 mg/dL | 0 | 2 | 0 | 2
Renal history [Number; unit: participants] — Moderately impaired = measured creatinine clearance (mCLcr) 30-59 mL/min, mildly impaired = mCLcr 60-89 mL/min, and normal = mCLcr ≥90 mL/min.
  participants
    Moderately impaired | 0 | 0 | 0 | 0
    Mildly impaired | 2 | 0 | 1 | 3
    Normal | 31 | 33 | 32 | 96
24-hour urine uric acid [Mean (Standard Deviation); unit: mg/24 hours] | 1000.6 (223.99) | 948.1 (231.16) | 909.4 (166.43) | 952.7 (210.44)
24-hour urine uric acid categories [Number; unit: participants] — Categories are based on tertiles, T1: 33.3rd percentile and T2: 66.6th percentile.
  participants
    ≤820 mg/24 hours (T1) | 9 | 13 | 11 | 33
    >820 to ≤987 mg/24 hours | 9 | 9 | 14 | 32
    >987 mg/24 hours (T2) | 15 | 11 | 8 | 34
24-hour urinary calcium [Mean (Standard Deviation); unit: mg/24 hours] | 240.1 (84.08) | 297.9 (77.60) | 278.7 (99.62) | 272.2 (90.00)
Lifetime kidney stone episodes [Mean (Standard Deviation); unit: kidney stone episodes] | 8.8 (10.18) | 12.5 (19.72) | 11.3 (14.97) | 10.9 (15.38)
Kidney stone passage [Number; unit: participants]
  No | 6 | 0 | 4 | 10
  Yes | 27 | 33 | 29 | 89
Composition of most recent passed stone [Number; unit: participants] — Includes participants with a kidney stone passage: 27, 33 and 29 participants for each treatment group, respectively.
  participants
    Calcium Oxalate | 8 | 14 | 13 | 35
    Uric acid | 1 | 0 | 0 | 1
    Calcium citrate | 0 | 0 | 1 | 1
    Unknown | 18 | 19 | 15 | 52
Kidney stone procedures [Number; unit: participants] — Participants may have had more than one kidney stone procedure.
  participants
    None | 13 | 13 | 18 | 44
    Shock Wave Lithotripsy | 17 | 20 | 14 | 51
    Ureteroscopy | 9 | 6 | 9 | 24
    Nephrolithotomy/Nephrolithotripsy | 3 | 2 | 0 | 5
    Open surgery | 2 | 2 | 2 | 6
    Other procedure | 2 | 4 | 2 | 8
    Stone Procedure | 20 | 20 | 15 | 55
Use of kidney stone drug [Number; unit: participants]
  None | 28 | 30 | 30 | 88
  Allopurinol | 2 | 1 | 0 | 3
  Other drug therapy | 3 | 2 | 3 | 8
Baseline in-plane Diameter of the largest Calcium Oxalate Stone [Mean (Standard Deviation); unit: mm] | 12.24 (7.363) | 9.34 (4.311) | 8.22 (3.756) | 9.91 (5.590)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Month 6 in 24-hour Urine Uric Acid (uUA) Excretion
Description: The change from Baseline to Month 6 in 24-hour urine uric acid is expressed as a percentage of the Baseline uUA value.
Time Frame: Baseline and Month 6
Population: The full analysis set (patients who took at least 1 dose of double-blind study drug and had a baseline 24-hour uUA >700 mg and at least 1 kidney CaOx stone ≥3 mm in its longest inplane diameter). Missing Month 6 values were imputed with baseline values if patient discontinued due to an AE; or otherwise with the last available post-baseline value.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Febuxostat | Allopurinol | Placebo
Number analyzed (Participants) | 33 | 33 | 33
percent change | -58.6 (28.56) | -36.4 (36.97) | -12.7 (28.81)
Statistical Analysis 1: Comparison: Febuxostat vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Hochberg's method for multiple comparisons was used to ensure that the overall 0.050 level of significance was maintained for comparisons of febuxostat to allopurinol and to placebo
Statistical Analysis 2: Comparison: Febuxostat vs Allopurinol; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percent Change From Baseline to Month 6 in the In-plane Diameter of the Largest Calcium Oxalate (CaOx) Stone
Description: Multidetector Computed Tomography (MDCT) was used to visualize and measure calcium oxalate kidney stones at Baseline and after 6 months of treatment. All MDCT images were analyzed independently by a Central Reader. The change from Baseline to month 6 is expressed as a percentage of the Baseline largest in-plane diameter.
Time Frame: Baseline and Month 6
Population: Full analysis set, for whom Baseline and Month 6 MDCT data were available. Measurements more than 1-day after a patient's last dose of study drug were not included.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Febuxostat | Allopurinol | Placebo
Number analyzed (Participants) | 27 | 24 | 29
percent change | -6.50 (28.357) | 0.63 (12.605) | 3.20 (23.697)
Statistical Analysis 1: Comparison: Febuxostat vs Placebo; Test type: Superiority or Other; p = 0.130, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat vs Allopurinol; Test type: Superiority or Other; p = 0.348, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline to Month 6 in the Number of Calcium Oxalate Stones
Description: Multidetector Computed Tomography (MDCT) was used to visualize and count calcium oxalate kidney stones at Baseline and after 6 months of treatment. All MDCT images were analyzed independently by a Central Reader.
Time Frame: Baseline and Month 6
Population: Full analysis set for whom both Baseline and Month 6 MDCT data were available. Measurements more than 1 day after a patient's last dose of study drug were not included.
Measure: Mean (Standard Deviation); unit: stones
Arm/Group | Febuxostat | Allopurinol | Placebo
Number analyzed (Participants) | 28 | 24 | 30
stones
  Baseline (n=28, 24, 30) | 4.84 (3.921) | 6.60 (6.832) | 5.57 (5.785)
  Change from Baseline (n=26, 23, 26) | -0.06 (1.602) | 0.28 (1.953) | 0.10 (1.817)
Statistical Analysis 1: Comparison: Febuxostat vs Placebo; Test type: Superiority or Other; p = 0.403, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat vs Allopurinol; Test type: Superiority or Other; p = 0.413, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline to Month 6 in 24-hour Measured Creatinine Clearance
Description: Creatinine clearance is a measure of how well the kidneys are filtering creatinine, a waste product produced by the muscles. Measured creatinine clearance was calculated according to the following: Urine 24 hour Creatinine/Serum Creatinine x (total Urine volume/elapsed time) x (1.73/body surface area).
Time Frame: Baseline and Month 6
Population: Full analysis set. Missing Month 6 Visit 24-hour mCLcr values are imputed by Month 3 values if the Month 3 value was available otherwise the patient was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m²
Arm/Group | Febuxostat | Allopurinol | Placebo
Number analyzed (Participants) | 33 | 33 | 33
mL/min/1.73m²
  Baseline (n=33, 33, 33) | 146.9 (57.88) | 146.0 (44.32) | 147.1 (53.46)
  Change from Baseline (n=30, 29, 30) | -9.0 (60.82) | -7.7 (83.28) | -19.0 (45.72)
Statistical Analysis 1: Comparison: Febuxostat vs Placebo; Test type: Superiority or Other; p = 0.5535, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-values are from ANOVA with treatment as a fixed effect
Statistical Analysis 2: Comparison: Febuxostat vs Allopurinol; Test type: Superiority or Other; p = 0.9400, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-values are from ANOVA with treatment as a fixed effect

ADVERSE EVENTS:
Time Frame: Treatment emergent AEs were defined as any AE, regardless of relationship to study drug, which occurred on or after the first double blind dose date and up to 30 days after the last dose date of the double-blind study drug (up to 7 months).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Febuxostat | Allopurinol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 1/33
Other Adverse Events (participants affected / at risk) | 14/33 | 13/33 | 12/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat (N=33) | Allopurinol (N=33) | Placebo (N=33)
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat (N=33) | Allopurinol (N=33) | Placebo (N=33)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 3
Nephrolithiasis (Renal and urinary disorders) | 3 | 1 | 3
Headache (Nervous system disorders) | 0 | 3 | 3
Oedema peripheral (General disorders) | 1 | 3 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0
Creatinine urine increased (Investigations) | 2 | 0 | 0
Urine calcium increased (Investigations) | 2 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.